CLINICAL TRIAL: NCT05110807
Title: Phase I Clinical Study to Evaluate the Tolerability and Pharmacokinetics of TQB3617 Capsule in Patients With Advanced Malignant Tumors
Brief Title: A Clinical Study to Evaluate the Tolerability and Pharmacokinetics of TQB3617 Capsule in Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3617-I-01
Record Dates: First submitted 2021-11-04; First posted 2021-11-08 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3617 (Experimental): 0.1mg, once daily, was used as the initial dose, and the medication stage was divided into single administration and continuous administration stages. The single administration was given once, and the continuous administration stage was entered 7 days after drug withdrawal. The drug was administered continuously until the disease progressed.
  Interventions: Drug: TQB3617

INTERVENTIONS:
Drug: TQB3617 — TQB3617 is a BET inhibitor.

SUMMARY:
TQB3617 is a bromodomain and extra-terminal (BET) inhibitor that can competitively bind to bromodomains (BRDs) with Acetylated lysine(Kac) and block or partially block the role of KAc in subsequent gene transcription and regulation of chromatin structure, thereby playing an anti-tumor role.

ELIGIBILITY:
Inclusion Criteria:

* Aged: ≥18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Life expectancy ≥ 3 months.
* Patients with advanced malignancy tumor who have failed standard treatment or are unable to receive standard treatment or have no effective treatment.
* Female and male subjects should agree to use an adequate method of contraception starting with signing informed consent form (ICF) through 180 days after the last dose of study. The women of reproductive age who blood/urine results were positivetherapy before the first study drug is administered within less than 7 days.

Exclusion Criteria:

* Patients has had or is currently having other malignant tumors within 3 years.
* Patients have multiple factors that affect their oral medication (such as inability to swallow, chronic diarrhea, and intestinal obstruction).
* The patient had unmitigated toxic reactions due to any prior treatment.
* Patients underwent major surgical treatment, open biopsy, or significant traumatic injury within 4 weeks prior to the start of study treatment.
* Patients have long - term unhealed wounds or fractures.
* Patients were taking Cytochrome P450 3A4, Cytochrome P450 3A5, Cytochrome P450 2A6, Cytochrome P450 2D6 (CYP3A4, CYP3A5, CYP2A6,CYP2D6) inhibitors or inducers before oral medication.
* Patients who, in the investigator's judgment, have a comorbidity that seriously endangers patient safety or interferes with study completion, or who are considered unsuitable for inclusion for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 48 weeks
  The highest dose of a drug or treatment that does not cause unacceptable side effects.
Adverse events (AEs) and serious adverse events (SAEs) | Baseline up to 48 weeks
  The occurrence of all AEs and SAEs

SECONDARY OUTCOMES:
Time to reach maximum (peak) plasma concentration following drug administration（Tmax） | Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8,12, 24, 48, 72, 96, 120,168 hours after oral administration of a single drug delivery; 30 minutes, 1, 2, 3, 4, 6, 8,12, 24 hours of day 28; 30 minutes before oral administration on day 8, day 15, day 22, day 28.
  To characterize the pharmacokinetics of TQB3617 by assessment of time to reach maximum plasma concentration after single and multiple dosing
Maximum (peak) plasma drug concentration （Cmax） | Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8,12, 24, 48, 72, 96, 120,168 hours after oral administration of a single drug delivery; 30 minutes, 1, 2, 3, 4, 6, 8,12, 24 hours of day 28; 30 minutes before oral administration on day 8, day 15, day 22, day 28.
  Cmax is the maximum plasma concentration of TQB3617 or metabolite(s).
Elimination half-life (to be used in one-or non- compartmental model) （t1/2） | Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8,12, 24, 48, 72, 96, 120,168 hours, after oral administration of a single drug delivery.
  t1/2 is time it takes for the blood concentration of TQB3617 or metabolite(s) to drop by half.
Maximum (peak) steady-state plasma drug concentration during a dosage interval （Cmax,ss） | Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8,12, 24, 48, 72, 96, 120,168 hours after oral administration of a single drug delivery; 30 minutes, 1, 2, 3, 4, 6, 8,12, 24 hours of day 28; 30 minutes before oral administration on day 8, day 15, day 22, day 28.
  Maximum (peak) steady-state plasma drug concentration during a dosage interval
Minimum steady-state plasma drug concentration during a dosage interval （Css-min） | Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8,12, 24, 48, 72, 96, 120,168 hours after oral administration of a single drug delivery; 30 minutes, 1, 2, 3, 4, 6, 8,12, 24 hours of day 28; 30 minutes before oral administration on day 8, day 15, day 22, day 28.
  Minimum steady-state plasma drug concentration during a dosage interval
Concentration at the end of the dosing interval AUCtau,ss | Pre-dose, 30 minutes, 1, 2, 3, 4, 6, 8,12, 24, 48, 72, 96, 120,168 hours after oral administration of a single drug delivery; 30 minutes, 1, 2, 3, 4, 6, 8,12, 24 hours of day 28; 30 minutes before oral administration on day 8, day 15, day 22, day 28.
  To characterize the pharmacokinetics of TQB3617 by assessment of area the concentration at the end of the administration interval
Overall response rate (ORR) | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).
Progress Free Survival（PFS） | up to 96 weeks
  From the start of randomization to the first tumor progression or time of death.
Disease control rate（DCR） | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 96 weeks
  The time when the participants first achieved complete or partial remission to disease progression.
Overall Survival（OS） | assessed up to 100 months
  From date of first administration of test drug until the date of death from any cause，

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Cen, Guangzhou, Guangdong
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Zhang Y, Yin Q, Zhao B, Liu F, Li S, Cai J, Fang X, Bai B, Nie M, Zou Q, Ding D, Wang X, Zhu J, Yu D, Wang X, Zhang X, Wang L, Xia Y, Cai Q. TQB3617, a bromodomain and extra-terminal inhibitor, in patients with relapsed or refractory lymphoma: A multicenter, phase 1 trial. Med. 2026 Jan 9;7(1):100893. doi: 10.1016/j.medj.2025.100893. Epub 2025 Oct 27. PMID 41151587